CLINICAL TRIAL: NCT00340704
Title: An Uncontrolled, Open-label, Titration, Long-term Safety (up to 12 Months) and Efficacy Study of Tamsulosin Hydrochloride in Children With Neuropathic Bladder, With a Randomized Pharmacokinetic Sub-study Investigating Low, Medium and High Dose Ranges.
Brief Title: PK/PD, Long-term Safety and Efficacy of Tamsulosin Treatment in Children With Neurogenic Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 527.66
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Bladder, Neurogenic
Keywords: tamsulosin; pediatric; neurogenic bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Low dose group (Experimental)
  Interventions: Drug: tamsulosin hydrochloride
- 2. Medium dose group (Experimental)
  Interventions: Drug: tamsulosin hydrochloride
- 3. High dose group (Experimental)
  Interventions: Drug: tamsulosin hydrochloride

INTERVENTIONS:
Drug: tamsulosin hydrochloride — oral

SUMMARY:
Aims of this study is to characterize the pharmacokinetic/pharmacodynamic profile and evaluate the safety, efficacy and tolerability, of tamsulosin hydrochloride as treatment in children with a neuropathic bladder, over the course of 12 months of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic bladder secondary to known neurological disorder
* Elevated detrusor leak point pressures (LPP) ≥40 cm H2O confirmed by two measurements at baseline

Exclusion Criteria:

* Clinically significant abnormalities as determined by the investigator
* A history of relevant orthostatic hypotension, fainting spells or blackouts

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (19):
  - Birmingham, Alabama
  - Los Angeles, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - St Louis, Missouri
  - Buffalo, New York
  - Lake Success, New York
  - Tarrytown, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin
- Ghent, Belgium
- Brazil (2):
  - Santo André
  - São Paulo
- Canada (3):
  - Halifax
  - Montreal
  - Toronto
- Germany (5):
  - Berlin
  - Deggendorf
  - Essen
  - Hamburg
  - Mainz
- India (13):
  - Ahmedabad
  - Belagavi
  - Bengaluru
  - Hyderabaad
  - Kochi
  - Lucknow
  - Ludhiana
  - Manipal
  - Mumbai
  - Nadiād
  - Nagpur
  - New Delhi
  - Pune
- Italy (3):
  - Cagliari
  - Florence
  - Roma
- Mexico (2):
  - León
  - Puebla City
- Philippines (3):
  - Manila
  - Pasig
  - Quezon City
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Africa (5):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Pretoria
  - Roodepoort
- South Korea (4):
  - Gwangju
  - Incheon
  - Pusan
  - Seoul
- Spain (3):
  - Barcelona
  - Madrid
  - Málaga
- Chernivtsy, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial has 3 different Data base locks (DBLs) based on 3 separate populations PK/PD, Group D-Denovo & Group D-527.51 Rollover. For population PK/PD the DBL date was 18July2007, Group D-Denovo the DBL date was 23Jan2009 & Group D-527.51 Rollover the DBL date was 11Sep2009.
Pre-assignment Details: Three different Clinical trial reports were prepared based on 3 separate populations (PK/PD, Group D-Denovo & Group D-527.51). Group D-Denovo includes patients from PK Phase & additional subjects & Group D-527.51 Rollover includes patients who successfully completed tamsulosin HCl Study 527.51
Groups:
- Tamsulosin - Low Dose Level (PK Study): Subjects randomized to low dose level (0.001-0.002 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In PK study, all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight. Depending on the results of the Leak point pressure (LPP) results, subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.
  Subjects with body weight of 12.1-25.0 kg received low dose of 0.025 mg qd (once daily), body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - Medium Dose Level (PK Study): Subjects randomized to medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In PK study, all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight. Depending on the results of the LPP results, subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.
  Subjects with body weight of 12.1-25.0 kg received medium dose of 0.05 mg qd, body weight of 25.1-50.0 kg received medium dose of 0.1 mg qd with and body weight of 50.1-100.0 kg received medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (PK Study): Subjects randomized to high dose level(0.004-0.008mg/kg) of tamsulosin hydrochloride,dependent on a subject's body weight.
  In PK study,all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight.Depending on the results of the LPP,subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.
  Subjects with body weight of 12.1-25.0kg received high dose of 0.1mg qd,body weight of 25.1-50.0kg received high dose of 0.2mg qd & body weight of 50.1-100.0kg received high dose of 0.4mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - Low Dose Level (Group D-Denovo): Subjects received low dose level (0.001 - 0.002 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In Group D-Denovo, all subjects started the study at the low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study.
  Subjects with body weight of 12.1-25.0 kg received low dose of 0.025 mg qd, body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - Medium Dose Level (Group D-Denovo): Subjects who were titrated to medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In Group D-Denovo, all subjects started the study at the Low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study.
  Subjects with body weight of 9.0-12.0 kg received medium dose of 0.025 mg qd as their starting dose, body weight of 12.1-25.0 kg could have titrated to a medium dose of 0.05 mg qd, body weight of 25.1-50.0 kg could have titrated to a medium dose of 0.1 mg qd and body weight of 50.1-100.0 kg could have titrated to a medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (Group D-Denovo): Subjects titrated to high dose level (0.004-0.008 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight.
  In Group D-Denovo, all subjects started the study at the Low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study.
  Subjects with body weight of 9.0-12.0 kg received high dose of 0.05 mg qd, body weight of 12.1-25.0 kg received high dose of 0.1 mg qd, body weight of 25.1-50.0 kg received high dose of 0.2 mg qd & body weight of 50.1- 100.0 kg received high dose of 0.4 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - Low Dose Level (Group D-527.51 Rollover): Subjects received low dose level (0.001-0.002 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight.
  In Group D- 527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial (527.66). All subjects were to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that that the higher doses would provide some efficacy.
  Subjects with body weight of 12.1-25.0 kg received low dose of 0.025 mg qd, body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg qd received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - Medium Dose Level (Group D-527.51 Rollover): Subjects who were to receive medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight.
  In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial. All subjects were to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that the higher doses would provide some efficacy.
  Subjects with body weight of 9.0-12.0 kg received medium dose of 0.025 mg qd, body weight of 12.1-25.0 kg received medium dose of 0.05 mg qd, body weight of 25.1-50.0 kg received medium dose of 0.1 mg qd, body weight of 50.1-100.0 kg received medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (Group D-527.51 Rollover): Subjects titrated to high dose level (0.004-0.008 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight.
  In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial. All subjects had to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that the higher doses would provide some efficacy.
  Subjects with body weight of 9.0-12.0 kg received high dose of 0.05 mg, body weight of 12.1-25.0 kg received high dose of 0.1 mg, body weight of 25.1-50.0 kg received high dose of 0.2 mg, body weight of 50.1-100.0 kg received high dose of 0.4 mg by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
Period: PK Study
Arm/Group | Tamsulosin - Low Dose Level (PK Study) | Tamsulosin - Medium Dose Level (PK Study) | Tamsulosin - High Dose Level (PK Study) | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Started | 10 | 10 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 10 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Group D- Denovo & 527.51 Rollover Study
Arm/Group | Tamsulosin - Low Dose Level (PK Study) | Tamsulosin - Medium Dose Level (PK Study) | Tamsulosin - High Dose Level (PK Study) | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Started | 0 | 0 | 0 | 29 | 21 | 37 | 54 | 13 | 29
PK Study Subjects Entered Group D-Denovo | 0 | 0 | 0 | 7 | 5 | 18 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 27 | 16 | 30 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 2 | 5 | 7 | 53 | 12 | 29
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Other reason not defined above | 0 | 0 | 0 | 0 | 0 | 3 | 53 | 11 | 28

BASELINE CHARACTERISTICS:
Population: Treated Set: Includes all patients who are dispensed study medication and are documented to have taken at least one dose of treatment. In this study, some of the subjects are in multiple phases: PK and Group D-Denovo. Thus, the baseline characteristics are based on the unique subject entered into the study.
Groups:
- Tamsulosin - Low Dose Level (Group D-Denovo): Subjects received low dose level (0.001 - 0.002 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight. In Group D-Denovo, all subjects started the study at the low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study. Subjects with body weight of 12.1- 25.0 kg received low dose of 0.025 mg qd, body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (Group D-Denovo): Subjects titrated to high dose level (0.004-0.008 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight. In Group D-Denovo, all subjects started the study at the Low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study. Subjects with body weight of 9.0-12.0 kg received high dose of 0.05 mg qd, body weight of 12.1-25.0 kg received high dose of 0.1 mg qd, body weight of 25.1-50.0 kg received high dose of 0.2 mg qd & body weight of 50.1-100.0 kg received high dose of 0.4 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Total: Total of all reporting groups
Arm/Group | Tamsulosin - Low Dose Level (PK Study) | Tamsulosin - Medium Dose Level (PK Study) | Tamsulosin - High Dose Level (PK Study) | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 22 | 16 | 19 | 54 | 13 | 29 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.5) | 6.5 (2.6) | 8.8 (3.7) | 6.8 (3.4) | 6.3 (3.7) | 8.1 (3.8) | 8.1 (3.8) | 7.0 (3.4) | 8.3 (4.1) | 7.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 5 | 12 | 7 | 10 | 21 | 8 | 12 | 83
  Male | 5 | 7 | 5 | 10 | 9 | 9 | 33 | 5 | 17 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of LPP Responders for Group D-Denovo and Group D-527.51 Rollover
Description: Group D-Denovo: Leak point pressure (LPP) Response at(response defined as a subject who achieves an LPP pressure <40 cm H2O) at the end of treatment based on two confirmatory values. Group D-527.51 Rollover: Leak point pressure (LPP) Response at (response defined as a subject who achieves an LPP pressure <40 cm H2O) last value of the treatment based on two confirmatory values. The last value on treatment included any final value prior to discontinuation of treatment, regardless of the length of treatment. Detrusor leak point pressure (LPP) recorded in cm H2O which was obtained using a standard urodynamic technique, a cystometrogram. Descriptive statistics were used to assess this endpoint. This Outcome Measure was only pre-specified for Group D-Denovo and Group D-527.51 Rollover subjects, so results of these two groups are provided.
Time Frame: Group D-Denovo: Week 52. Group D-527.51 Rollover: Week 1, Week 2, Week 3 and Week 4 prior to dose administration and Week9 (optional), Week 13 (additional), Week 26 (optional) and Week 52 after drug administration.
Population: Full analysis set (FAS-LPP): This subject set includes all subjects in the Treated set who received one dose of treatment and had one on treatment LPP measurement.
Measure: Number; unit: percentage of responders
Groups:
- Tamsulosin - Medium Dose Level (Group D-527.51 Rollover): Subjects who were to receive medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight.
  In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial. All subjects were to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that the higher doses would provide some efficacy.
  Subjects with body weight of 9.0-12.0 kg received medium dose of 0.025 mg qd, body weight of 12.1-25.0 kg received medium dose of 0.05 mg qd , body weight of 25.1-50.0 kg received medium dose of 0.1 mg qd, body weight of 50.1-100.0 kg received medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
Arm/Group | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 26 | 14 | 30 | 53 | 12 | 29
percentage of responders | 73.1 | 35.7 | 26.7 | 67.9 | 58.3 | 20.7

2. Primary Outcome: Number of LPP Responders at Each Visit Over Time (Classified by Last Value on Treatment) for Group D-527.51 Rollover.
Description: Number of Leak point pressure (LPP) Responders at each visit (week) over time (classified by last value on treatment). Due to the early termination of the study, most of the LPP assessments were conducted within Weeks 1-9 of treatment. Summary of LPP response rates provided over time.The subjects are classified according to the treatment they were receiving at the last value on treatment. Therefore, no assumptions can be made regarding what dose they were receiving at a particular time point. LD: Low Dose, MD: Medium Dose and HD: High Dose This Outcome Measure was only pre-specified for Group D-527.51 Rollover subjects, so results of this group is provided.
Time Frame: Week 1 (Visit 3) , Week 2 (Visit 4) , Week 3 (Visit 5) and Week 4 (Visit 6) prior to dose administration and Week 9 (Visit 7) (optional), Week 13 (Visit 8) (additional), Week 26 (Visit 9) (optional) and Week 52 (Visit 11) after drug administration.
Population: Full analysis set (FAS-LPP)
Measure: Number; unit: Participants
Arm/Group | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 53 | 12 | 29
Participants
  Week 1 (N= 40 (LD), 12 (MD), 27 (HD)) | 38 | 1 | 0
  Week 2 (N= 2 (LD), 7 (MD), 27 (HD)) | 2 | 7 | 2
  Week 3 (N= 3 (LD), 0 (MD), 22 (HD)) | 2 | 0 | 5
  Week 4 (N= 1 (LD), 0 (MD), 3 (HD)) | 1 | 0 | 0
  Week 9 (N= 7 (LD), 2 (MD), 16 (HD)) | 5 | 2 | 5
  Week 13 (N= 4 (LD), 0 (MD), 2 (HD)) | 1 | 0 | 1
  Week 26 (N= 2 (LD), 0 (MD), 3 (HD)) | 1 | 0 | 1
  Week 52 (N= 1 (LD), 1 (MD), 0 (HD)) | 1 | 1 | 0

3. Secondary Outcome: Early Responders Who Maintained Their LPP Below 40 cm H2O During the Study for Group D-Denovo and Group D-527.51 Rollover
Description: Early responders who maintained their detrusor leak point pressure (LPP) below 40 cm H2O during the study. Timeframe for Group D-Denovo: Low dose: Week 1, 3 & 4 prior to dose and Week 2, 9 & 26 (optional), 13(additional) & 52 post dose. Medium dose: Week 1, 2 & 4 prior to dose and Week 3, 9(optional), 13(additional), 26 (optional) & 52 post dose. High dose: Week 1, 2 & 3 prior to dose administration and Week 4, 9(optional), 13(additional), 26 (optional) & 52 post dose. Group D-527.51 Rollover: Week 1, 2,3 & 4 prior to dose and Week 9 &26 (optional),13 (additional) & 52 post dose. This Outcome Measure was only pre-specified for Group D-Denovo and Group D-527.51 Rollover subjects, However this endpoint was not analysed for Group D-527.51 Rollover as very limited data were collected due to early termination of the study & no alternative endpoint was defined in the Group D-527.51 rollover, so only the results for Group D-Denovo is provided.
Time Frame: Week 1 to Week 52 (Time frame for all weeks are described study wise in the Description).
Population: Full analysis set (FAS-LPP)
Measure: Number; unit: Participants
Groups:
- Tamsulosin-low Dose Level (Group D-Denovo): Subjects received low dose level (0.001 - 0.002 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In Group D-Denovo, all subjects started the study at the low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study.
  Subjects with body weight of 12.1- 25.0 kg received low dose of 0.025 mg qd, body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin-medium Dose Level (Group D-Denovo): Subjects who were titrated to medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In Group D-Denovo, all subjects started the study at the Low Dose level, with the exception of the children with a body weight between 9 kg and 12 kg (they started at the Medium Dose level), and titrated up to higher dose levels on a weekly basis until an efficacious level was reached. The subjects remained on their efficacious dose level for the remainder of the study.
  Subjects with body weight of 9.0-12.0 kg received medium dose of 0.025 mg qd as their starting dose, body weight of 12.1-25.0 kg could have titrated to a medium dose of 0.05 mg qd, body weight of 25.1-50.0 kg could have titrated to a medium dose of 0.1 mg qd and body weight of 50.1-100.0 kg could have titrated to a medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
Arm/Group | Tamsulosin-low Dose Level (Group D-Denovo) | Tamsulosin-medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 28 | 21 | 37 | 0 | 0 | 0
Participants | 17 | 5 | 3 |  |  |

4. Secondary Outcome: Change From Baseline in LPP for Group D-527.51 Rollover
Description: Median change from baseline in detrusor leak point pressure (LPP) by treatment group (subjects are classified according to the treatment they were taking at end of treatment) and week. Baseline assessments were obtained from trial 527.51 for Group D-527.51 Rollover. The results from Week 1 were reported because there were very few subjects who reported data at subsequent visits due to the termination of the trial. This Outcome Measure was only pre-specified for Group D-527.51 Rollover subjects, so results of this group is provided.
Time Frame: Baseline and week 1
Population: Full analysis set (FAS-LPP)
Measure: Median (Standard Deviation); unit: cm H2O
Arm/Group | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 53 | 12 | 29
cm H2O
  Baseline (N= 53 (LD), 12 (MD), 29(HD)) | 48.50 (14.47) | 48.5 (11.19) | 55.50 (24.52)
  Week 1 - Actual (N= 39 (LD), 9 (MD),22 (HD)) | 29.00 (8.50) | 49.50 (8.30) | 64.75 (27.20)
  Week 1 - Change (N= 39 (LD), 9 (MD),22 (HD)) | -25.5 (15.18) | -2 (13.68) | -1.25 (24.97)

5. Secondary Outcome: Percent Change From Baseline in LPP for Group D-527.51 Rollover
Description: Percent change from baseline in actual detrusor leak point pressure (LPP) by treatment group (subjects are classified according to the treatment they were taking at end of treatment) and Week. Baseline assessments were obtained from trial 527.51 for Group D-527.51 Rollover. The results from Week 1 were reported because there were very few subjects who reported data at subsequent visits due to the termination of the trial. This Outcome Measure was only pre-specified for Group D-527.51 Rollover subjects, so results of this group is provided.
Time Frame: Baseline and Week 1
Population: Full analysis set (FAS-LPP)
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 53 | 12 | 29
percent change
  Baseline (N= 53 (LD), 12 (MD), 29 (HD)) | 48.50 (14.47) | 48.50 (11.19) | 55.50 (24.52)
  Week 1 - Actual (N= 39 (LD), 9 (MD), 22 (HD)) | 29.00 (8.50) | 49.50 (8.30) | 64.75 (27.20)
  Week 1 - Change (N= 39 (LD), 9 (MD), 22 (HD)) | -48.48 (18.65) | -3.88 (22.43) | -2.71 (40.41)

6. Secondary Outcome: Response Defined as Stabilization or Improvement of Hydroureter Measured by Renal Ultrasound Compared to Baseline for Group D-Denovo and Group D-527.51 Rollover
Description: Response defined as stabilization or improvement of hydroureter measured by renal ultrasound compared to baseline by treatment group (subjects are classified according to the treatment they were taking at Week 52 or end of treatment) at week 52 for Group D-Denovo and (subjects are classified according to the treatment they were taking at the end of treatment) at last value on treatment for Group D-527.51 Rollover. Baseline assessments were obtained from trial 527.51 for Group D-527.51 Rollover. The overall treatment duration was not sufficient to reach any meaningful conclusions regarding improvement or stabilization of hydroureter in the Group D-527.51 Rollover. Hydroureter response is defined as improvement or stabilization based upon the presence or absence of hydroureter at end of treatment compared to baseline. This Outcome Measure was only pre-specified for Group D-Denovo and Group D-527.51 Rollover subjects, so results of these two groups are provided.
Time Frame: Group D-Denovo: Baseline and Week 52. Group D-527.51 Rollover: Baseline, Week 26 and Week 52.
Population: Full analysis set (FAS-RENAL): Includes all patients in the Treated set who received one dose of treatment and had one on treatment renal measurement.
Measure: Number; unit: Participants
Arm/Group | Tamsulosin-low Dose Level (Group D-Denovo) | Tamsulosin-medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 27 | 17 | 34 | 44 | 8 | 19
Participants
  Right Kidney | 26 | 15 | 28 | 43 | 8 | 19
  Left Kidney | 24 | 14 | 29 | 43 | 8 | 17

7. Secondary Outcome: Response Defined as Stabilization or Improvement of Hydronephrosis Measured by Renal Ultrasound Compared to Baseline for Group D-Denovo and Group D-527.51 Rollover
Description: Response defined as stabilization or improvement of hydronephrosis measured by renal ultrasound compared to baseline by treatment group (subjects are classified according to the treatment they were taking at Week 52 or end of treatment) at week 52 for Group D-Denovo and (subjects are classified according to the treatment they were taking at the end of treatment) at last value on treatment for Group D-527.51 Rollover. Baseline assessments were obtained from trial 527.51 for Group D-527.51 Rollover. The overall treatment duration was not sufficient to reach any meaningful conclusions regarding improvement or stabilization of hydronephrosis in the Group D-527.51 Rollover. Hydronephrosis response is defined as an improvement or stabilization based upon ultrasound grading at the end of the study. The lower or same grade at end of treatment compared to baseline is considered an improvement or stabilization.
Time Frame: Group D-Denovo: Baseline and Week 52. Group D-527.51 Rollover: Baseline, Week 26 and Week 52.
Population: Full analysis set (FAS-RENAL). This Outcome Measure was only pre-specified for Group D-Denovo and Group D-527.51 Rollover subjects, so results of these two groups are provided.
Measure: Number; unit: Participants
Arm/Group | Tamsulosin-low Dose Level (Group D-Denovo) | Tamsulosin-medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 27 | 17 | 34 | 44 | 8 | 19
Participants
  Right Kidney | 26 | 15 | 28 | 39 | 8 | 17
  Left Kidney | 24 | 14 | 26 | 42 | 7 | 17

8. Secondary Outcome: LPP Response at Any Time During the Trial for Group D-Denovo and Group D-527.51 Rollover
Description: Response rates of LPP responders (2 LPP values < 40 cm H2O) at any time during the trial by treatment group. Timeframe for Group D-Denovo: Low dose: Week 1, 3 & 4 prior to dose and Week 2, 9 & 26 (optional), 13(additional) & 52 post dose. Medium dose: Week 1, 2 & 4 prior to dose and Week 3, 9(optional), 13(additional), 26 (optional) & 52 post dose. High dose: Week 1, 2 & 3 prior to dose administration and Week 4, 9(optional), 13(additional), 26 (optional) & 52 post dose. Group D-527.51 Rollover: Week 1, 2, 3 & 4 prior to dose and Week 9 &26 (optional),13 (additional) & 52 post dose. This Outcome Measure was only pre-specified for Group D-Denovo and Group D-527.51 Rollover subjects, so results of these two groups are provided.
Time Frame: Week 1 to Week 52 (described study wise in the Description).
Population: Full analysis set (FAS-LPP)
Measure: Number; unit: participants
Arm/Group | Tamsulosin-low Dose Level (Group D-Denovo) | Tamsulosin-medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 28 | 21 | 37 | 53 | 12 | 29
participants | 26 | 16 | 16 | 42 | 8 | 12

9. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic Testing, Electrocardiogram (ECG), Laboratory Values,Urinalysis,Occurence of Adverse Events & Cognitive Testing for Group D-527.51 Rollover
Description: Number of participants with Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic testing, Electrocardiogram (ECG), Laboratory Values, Urinalysis, Occurence of Adverse events and Cognitive Testing. Relevant findings or worsening of baseline conditions were reported as adverse events. Below mentioned result are the number of subjects who had the clinical relevant abnormalities for the preferred term 'Hepatic enzyme increased'. This Outcome Measure was only pre-specified for Group D-527.51 Rollover subjects, so results of this group is provided.
Time Frame: From first drug administration until 28 days after last study drug administration, upto 395 days
Population: Treated Set (TS)
Measure: Number; unit: Participants
Arm/Group | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 54 | 13 | 29
Participants | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic Testing, Electrocardiogram (ECG), Laboratory Values, Urinalysis, Occurence of Adverse Events and Cognitive Testing for Group D-Denovo
Description: Number of participants with Clinically Relevant Abnormalities for Physical Examination, Vital Signs/Orthostatic testing, Electrocardiogram (ECG), Laboratory Values, Urinalysis, Occurence of Adverse events and Cognitive Testing. Relevant findings or worsening of baseline conditions were reported as adverse events. Subjects who experienced orthostatic hypotension during orthostatic testing were reported as adverse events. This Outcome Measure was only pre-specified for Group D-Denovo, so results of this group is provided.
Time Frame: From first drug administration until 28 days after last study drug administration, upto 450 days
Population: Treated Set (TS)
Measure: Number; unit: Participants
Arm/Group | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo)
Number analyzed (Participants) | 29 | 21 | 37
Participants
  Blood urine present | 0 | 0 | 1
  Body temperature increased | 0 | 0 | 1
  Orthostatic hypotension | 1 | 3 | 0

11. Secondary Outcome: Vision Testing for Group D-Denovo
Description: Number of subjects with a change from baseline in visual acuity by treatment group (subjects are classified according to the treatment they were taking at Week 52 or end of treatment). They were analysed based on the below mentioned category in both the Eyes: 1) No Change 2) Decrease in visual acuity 3) Increase in visual acuity 4) Missing. Missing includes subjects with no baseline exam and subjects with exam scores missing. This Outcome Measure was only pre-specified for Group D-Denovo subjects, so results of this group is provided.
Time Frame: Baseline, Week 26 and Week 52.
Population: Treated Set (TS)
Measure: Number; unit: Participants
Arm/Group | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo)
Number analyzed (Participants) | 29 | 21 | 37
Participants
  Right Eye (Week 26) - No Change | 11 | 7 | 12
  Right Eye (Week 26) - Decrease in visual acuity | 8 | 1 | 8
  Right Eye (Week 26) - Increase in visual acuity | 8 | 4 | 11
  Right Eye (Week 26) - Missing | 2 | 9 | 6
  Left Eye (Week 26) - No Change | 11 | 6 | 19
  Left Eye (Week 26) - Decrease in visual acuity | 7 | 1 | 4
  Left Eye (Week 26) - Increase in visual acuity | 9 | 5 | 8
  Left Eye (Week 26) - Missing | 2 | 9 | 6
  Right Eye (Week 52) - No Change | 7 | 6 | 16
  Right Eye (Week 52) - Decrease in visual acuity | 10 | 2 | 4
  Right Eye (Week 52) - Increase in visual acuity | 11 | 6 | 12
  Right Eye (Week 52) - Missing | 1 | 7 | 5
  Left Eye (Week 52) - No Change | 11 | 5 | 12
  Left Eye (Week 52) - Decrease in visual acuity | 6 | 3 | 6
  Left Eye (Week 52) - Increase in visual acuity | 11 | 7 | 14
  Left Eye (Week 52) - Missing | 1 | 6 | 5

12. Secondary Outcome: Vision Testing for Group D-527.51 Rollover
Description: Number of subjects with a change from baseline in visual acuity by treatment group (subjects are classified according to the treatment they were taking at end of treatment). They were analysed based on the below mentioned category in both the Eyes: 1) No Change 2) Decrease in visual acuity 3) Increase in visual acuity 4) Missing. Missing includes subjects with no baseline exam and subjects with exam scores missing. This Outcome Measure was only pre-specified for Group D-527.51 Rollover subjects, so results of this group is provided.
Time Frame: Baseline and Week 52
Population: Treated Set (TS)
Measure: Number; unit: Participants
Arm/Group | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Number analyzed (Participants) | 54 | 13 | 29
Participants
  Right Eye - No Change | 32 | 10 | 12
  Right Eye - Decrease in visual acuity | 5 | 2 | 4
  Right Eye - Increase in visual acuity | 12 | 1 | 6
  Right Eye - Missing | 5 | 0 | 7
  Left Eye - No Change | 31 | 12 | 12
  Left Eye - Decrease in visual acuity | 8 | 1 | 3
  Left Eye - Increase in visual acuity | 10 | 0 | 7
  Left Eye - Missing | 5 | 0 | 7

13. Secondary Outcome: Cmax,1
Description: Maximum measured concentration of the analyte in plasma following the first dose, Cmax,1. This Outcome Measure was only pre-specified for PK Study- single dose group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h and 8h after the drug administration.
Population: Pharmacokinetics single dose set (PK-SD): This set includes subjects who were randomized, successfully took and retained the first dose of study medication and provided blood samples for PK at Visit 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK Study - Single Dose: Subjects received low dose level (0.001 - 0.002 mg/kg) of tamsulosin hydrochloride once daily dependent on a subject's body weight (12.1 - 25.0 kg, 25.1 - 50.0 kg and 50.1 - 100.0 kg), by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
  In PK Single dose study, it was planned to obtain the Low dose PK data after single dose from all the 30 patients randomized to Low, Medium and high. However as per the protocol amendment, the PK sampling after first drug administration of low dose level was stopped after inclusion of 11 patients and therefore the PK sample of 11 patients were evaluated for PK single dose.
Arm/Group | PK Study - Single Dose
Number analyzed (Participants) | 11
ng/mL | 1.67 (68.80)

14. Secondary Outcome: Tmax, 1
Description: Time from dosing to maximum measured concentration of the analyte in plasma after administration of the first dose, tmax, 1. This Outcome Measure was only pre-specified for PK Study- single dose group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h and 8h after the drug administration.
Population: Pharmacokinetics single dose set (PK-SD)
Measure: Median (Full Range); unit: hours
Arm/Group | PK Study - Single Dose
Number analyzed (Participants) | 11
hours | 6 [2 to 8]

15. Secondary Outcome: Cmax, 1 ,DW ,Norm
Description: Dose- and weight-normalized Cmax,1 (Cmax,1,DW,norm). Weight normalization of Cmax,1 was performed by dividing the respective quantities by the reciprocal of body weight in kg. This Outcome Measure was only pre-specified for PK Study- single dose group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h and 8h after the drug administration.
Population: Pharmacokinetics single dose set (PK-SD)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg*kg
Arm/Group | PK Study - Single Dose
Number analyzed (Participants) | 11
ng/mL/mg*kg | 1120 (67.20)

16. Secondary Outcome: Cpre,ss
Description: Pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose, Cpre,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS): This set includes subjects who were randomized successfully took study medication for two weeks at their randomized dose level and provided blood samples for PK at their steady state visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Tamsulosin - Low Dose Level (Steady State - PK Study): Subjects randomized to low dose level (0.001-0.002 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In PK study, all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight. Depending on the results of the Leak point pressure (LPP) results, subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.
  Subjects with body weight of 12.1-25.0 kg received low dose of 0.025 mg qd (once daily), body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - Medium Dose Level (Steady State - PK Study): Subjects randomized to medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight.
  In PK study, all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight. Depending on the results of the LPP results, subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.
  Subjects with body weight of 12.1-25.0 kg received medium dose of 0.05 mg qd, body weight of 25.1-50.0 kg received medium dose of 0.1 mg qd with and body weight of 50.1-100.0 kg received medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (Steady State - PK Study): Subjects randomized to high dose level(0.004-0.008mg/kg) of tamsulosin hydrochloride,dependent on a subject's body weight.In PK study,all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight.Depending on the results of the LPP,subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy.Subjects with body weight of 12.1-25.0kg received high dose of 0.1mg qd, body weight of 25.1-50.0kg received high dose of 0.2mg qd & body weight of 50.1-100.0kg received high dose of 0.4mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.One subject randomised to high dose level was not treated. Although actual number of subjects started is 11,10 were reported to ensure consistent reporting with baseline characteristics that includes only treated subjects.
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 9 | 9 | 10
ng/mL | 0.914 (159) | 1.83 (131) | 4.03 (70.60)

17. Secondary Outcome: Cmax,ss
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ, Cmax,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
ng/mL | 2.79 (59.50) | 5.02 (94.80) | 14.10 (50.30)
Statistical Analysis 1: Comparison: Tamsulosin - Low Dose Level (Steady State - PK Study) vs Tamsulosin - Medium Dose Level (Steady State - PK Study) vs Tamsulosin - High Dose Level (Steady State - PK Study); Dose proportionality for Cmax,ss was explored based on the regression model; Test type: Superiority or Other; Slope = 1.0039, 95% CI [0.6499 to 1.3579], Standard Error of Mean 0.1725 — Based on the estimate for the slope parameter, a two sided 95% confidence interval for the slope was computed. Perfect dose proportionality would correspond to a slope of 1. Standard error (SE) of the mean is actually SE of the slope

18. Secondary Outcome: Cmax,ss, DW, Norm
Description: Dose- and weight-normalized for Cmax,ss, Cmax,ss, DW, norm. Weight normalization of Cmax,ss was performed by dividing the respective quantities by the reciprocal of body weight in kg. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg*kg
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
ng/mL/mg*kg | 2040 (74.30) | 1850 (85.70) | 2240 (47.60)

19. Secondary Outcome: Cmin,ss
Description: Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ, Cmin,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
ng/mL | 0.747 (99.70) | 1.52 (130) | 4.01 (68.50)

20. Secondary Outcome: Tmax,ss
Description: Time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ, tmax,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Median (Full Range); unit: hours
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
hours | 5.00 (99.7) [2.33 to 8.00] | 5.92 (130) [2.00 to 8.00] | 5.01 (68.5) [2.23 to 8.00]

21. Secondary Outcome: AUCτ,ss
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ , AUCτ,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
ng*h/mL | 35.80 (75.60) | 68.20 (94.70) | 175.00 (61.00)
Statistical Analysis 1: Comparison: Tamsulosin - Low Dose Level (Steady State - PK Study) vs Tamsulosin - Medium Dose Level (Steady State - PK Study) vs Tamsulosin - High Dose Level (Steady State - PK Study); Dose proportionality for AUCτ,ss was explored based on the regression model; Test type: Superiority or Other; Slope = 0.98, 95% CI [0.5934 to 1.3666], Standard Error of Mean 0.1884 — Based on the estimate for the slope parameter, a two sided 95% confidence interval for the slope was computed. Perfect dose proportionality would correspond to a slope of 1. Standard error of the mean is actually standard error of the slope

22. Secondary Outcome: AUCτ ,ss ,DW ,Norm
Description: Dose- and weight-normalized of AUCτ ,ss ( AUCτ ,ss ,DW ,norm). Weight normalization of AUCτ,ss was performed by dividing the respective quantities by the reciprocal of body weight in kg. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg*kg
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
ng*h/mL/mg*kg | 26100 (91.10) | 25200 (82.90) | 27700 (59.10)

23. Secondary Outcome: λz,ss
Description: Terminal rate constant of the analyte in plasma at steady state, λz,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hours
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
1/hours | 0.0589 (48.10) | 0.0671 (40.80) | 0.0496 (31.90)

24. Secondary Outcome: t1/2,ss
Description: Terminal half-life of the analyte in plasma at steady state, t1/2,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
hours | 11.80 (48.10) | 10.30 (40.80) | 14.00 (31.90)

25. Secondary Outcome: MRTpo,ss
Description: Mean residence time of the analyte in the body at steady state after oral administration,MRTpo,ss. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
hours | 18.70 (50.50) | 17.60 (35.00) | 20.90 (23.60)

26. Secondary Outcome: CL/F,ss,W,Norm
Description: Weight-normalized CL/F,ss (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration), CL/F,ss,W,norm. Weight-normalized CL/F,ss was calculated by dividing the respective quantities by body weight in kg. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
L/h/kg | 0.0383 (91.10) | 0.0397 (82.90) | 0.0361 (59.10)

27. Secondary Outcome: Vz/F,ss,W,Norm
Description: Weight-normalized Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration), Vz/F,ss,W,norm. Weight-normalized VzF,ss was calculated by dividing the respective quantities by body weight in kg. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results of this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 10 | 9 | 10
L/kg | 0.65 (83.80) | 0.591 (103.00) | 0.729 (96.00)

28. Secondary Outcome: RA,Cmax
Description: The accumulation ratio was calculated from the patients who were randomised to the low dose group and for whom both parameters at first dose and steady state dose were available. Accumulation ratios of tamsulosin HCl in plasma at steady state after multiple dose administration over a uniform dosing interval τ, expressed as ratio of Cmax at steady state and after single dose. The accumulation ratio RA,Cmax was calculated as: Cmax,ss/Cmax,1. This Outcome Measure was only pre-specified for PK Study- steady state group subjects, so results from this group is provided.
Time Frame: -0.25h prior to dose and 2h, 4h, 6h, 8h, 10h, 24h and 33h after the drug administration.
Population: Pharmacokinetics steady state set (PK-SS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study)
Number analyzed (Participants) | 4
Ratio | 1.58 (65.20)

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last study drug administration, upto 80 days (Steady State - PK study), upto 450 days (Group D-Denovo) and upto 395 days (Group D-527.51 Rollover).
Description: Subjects were titrated to their efficacious dose.Based on LPP results,subjects could remain on that dose if it was found to be efficacious or titrate up to their higher doses which might have provided some efficacy.Therefore some of the subjects were counted more than once for having reported adverse events with different doses of the study.
Groups:
- Tamsulosin - High Dose Level (Steady State - PK Study): Subjects randomized to high dose level(0.004-0.008mg/kg) of tamsulosin hydrochloride, dependent on a subject's body weight. In PK study,all subjects were titrated to their randomized dose level that they needed to receive which was based on their weight. Depending on the results of the LPP,subjects could remain on that dose if it was found to be efficacious or go back to a lower efficacious dose or titrate up in hopes that the higher dose would provide some efficacy. Subjects with body weight of 12.1-25.0kg received high dose of 0.1mg qd, body weight of 25.1-50.0kg received high dose of 0.2mg qd & body weight of 50.1-100.0kg received high dose of 0.4mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - Low Dose Level (Group D-527.51 Rollover): Subjects received low dose level (0.001-0.002 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight. In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial (527.66). All subjects were to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that that the higher doses would provide some efficacy. Subjects with body weight of 12.1-25.0 kg received low dose of 0.025 mg qd, body weight of 25.1-50.0 kg received low dose of 0.05 mg qd and body weight of 50.1-100.0 kg qd received low dose of 0.1 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt, taken 30 minutes after breakfast.
- Tamsulosin - Medium Dose Level (Group D-527.51 Rollover): Subjects who were to receive medium dose level (0.002-0.004 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight. In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial. All subjects were to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that the higher doses would provide some efficacy. Subjects with body weight of 12.1-25.0 kg received low dose of 0.05 mg qd, body weight of 25.1-50.0 kg received medium dose of 0.1 mg qd, body weight of 50.1-100.0 kg received medium dose of 0.2 mg qd by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
- Tamsulosin - High Dose Level (Group D-527.51 Rollover): Subjects titrated to high dose level (0.004-0.008 mg/kg) of tamsulosin hydrochloride, once daily dependent on a subject's body weight. In Group D-527.51 Rollover, once subjects exited the double-blind trial they were rolled over into this trial. All subjects had to titrate to their efficacious dose. Doses that were available were based on subject's weight. Depending on the LPP results, subjects could remain on that dose if it was found to be efficacious or titrate up in hopes that the higher doses would provide some efficacy. Subjects with body weight of 12.1-25.0 kg received high dose of 0.1 mg, body weight of 25.1-50.0 kg received high dose of 0.2 mg, body weight of 50.1-100.0 kg received high dose of 0.4 mg by sprinkling the content of the capsule(s) over teaspoon of apple sauce or yogurt taken 30 minutes after breakfast.
Arm/Group | Tamsulosin - Low Dose Level (Steady State - PK Study) | Tamsulosin - Medium Dose Level (Steady State - PK Study) | Tamsulosin - High Dose Level (Steady State - PK Study) | Tamsulosin - Low Dose Level (Group D-Denovo) | Tamsulosin - Medium Dose Level (Group D-Denovo) | Tamsulosin - High Dose Level (Group D-Denovo) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) | Tamsulosin - High Dose Level (Group D-527.51 Rollover)
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10 | 2/82 | 3/61 | 4/41 | 1/93 | 1/41 | 1/29
Other Adverse Events (participants affected / at risk) | 5/10 | 5/10 | 3/10 | 51/82 | 25/61 | 33/41 | 31/93 | 10/41 | 9/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamsulosin - Low Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - Medium Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - High Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - Low Dose Level (Group D-Denovo) (N=82) | Tamsulosin - Medium Dose Level (Group D-Denovo) (N=61) | Tamsulosin - High Dose Level (Group D-Denovo) (N=41) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) (N=93) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) (N=41) | Tamsulosin - High Dose Level (Group D-527.51 Rollover) (N=29)
Tibial torsion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritoneal cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Tethered cord syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tamsulosin - Low Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - Medium Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - High Dose Level (Steady State - PK Study) (N=10) | Tamsulosin - Low Dose Level (Group D-Denovo) (N=82) | Tamsulosin - Medium Dose Level (Group D-Denovo) (N=61) | Tamsulosin - High Dose Level (Group D-Denovo) (N=41) | Tamsulosin - Low Dose Level (Group D-527.51 Rollover) (N=93) | Tamsulosin - Medium Dose Level (Group D-527.51 Rollover) (N=41) | Tamsulosin - High Dose Level (Group D-527.51 Rollover) (N=29)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 2 | 2 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 9 | 4 | 3 | 3 | 2 | 0
Catheter related complication (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 12 | 3 | 6 | 1 | 1 | 1
Suprapubic pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 1 | 5 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 4 | 3 | 1 | 5 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 11 | 1 | 2 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 15 | 11 | 16 | 9 | 3 | 4
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 8 | 2 | 3 | 2 | 1 | 2
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 7 | 1 | 3 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
In Group D-527.51 Rollover study, due to the early termination caution should be used in interpreting these results due to the impact of the early termination, as well as the impact of the study design on interpretation of results by dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.